CLINICAL TRIAL: NCT04485884
Title: An Open-label, Randomized, Single and Multiple Dosing Phase I Clinical Trial to Evaluate Pharmacokinetics/Pharmacodynamics and Safety/Tolerability of IN-C005 After Oral Administration in Healthy Korean and Caucasian Male Subjects
Brief Title: A Study to Evaluate Pharmacokinetics/Pharmacodynamics and Safety/Tolerability of IN-C005 in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IN_BTK_101
Record Dates: First submitted 2020-07-15; First posted 2020-07-24 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental): IN-C005 dose A
  Interventions: Drug: IN-C005 dose A
- Group B (Experimental): IN-C005 dose B
  Interventions: Drug: IN-C005 dose B
- Group C (Experimental): IN-C005 dose C
  Interventions: Drug: IN-C005 dose C
- Group D (Experimental): IN-C005 dose D
  Interventions: Drug: IN-C005 dose D
- Group E (Experimental): IN-C005 dose E
  Interventions: Drug: IN-C005 dose E
- Group F (Experimental): IN-C005 dose F
  Interventions: Drug: IN-C005 dose F

INTERVENTIONS:
Drug: IN-C005 dose A — One time dose of IN-C005 dose A taken orally.
  Other Names: IN-C005
  Arms: Group A
Drug: IN-C005 dose B — One time dose of IN-C005 dose B taken orally.
  Other Names: IN-C005
  Arms: Group B
Drug: IN-C005 dose C — One time dose of IN-C005 dose C taken orally.
  Other Names: IN-C005
  Arms: Group C
Drug: IN-C005 dose D — Oral administration of IN-C005 dose D once daily for 7 days.
  Other Names: IN-C005
  Arms: Group D
Drug: IN-C005 dose E — Oral administration of IN-C005 dose E once daily for 7 days.
  Other Names: IN-C005
  Arms: Group E
Drug: IN-C005 dose F — Oral administration of IN-C005 dose F once daily for 7 days.
  Other Names: IN-C005
  Arms: Group F

SUMMARY:
The main purpose of this study is to evaluate pharmacokinetics/pharmacodynamics and safety/tolerability of IN-C005 after oral administration in healthy Korean and Caucasian male subjects.

DETAILED DESCRIPTION:
[Pharmacokinetic Assessments]: Plasma concentrations of IN-C005 and its metabolite will be measured

1. Single Dosing Group (Korean Subjects)

   * Primary endpoints: Cmax and AUClast of IN-C005
   * Secondary endpoints: AUClast, Cmax, AUCinf, Tmax, t½, CL/F, and Vd/F of M1; AUCinf, Tmax, t½, CL/F, and Vd/F of IN-C005
2. Multiple Dosing Group (Caucasian Subjects)

   * Primary endpoints: Cmax, AUClast, Cmax,ss, and AUCτ,ss of IN-C005
   * Secondary endpoints: For M1, AUClast, Cmax, Cmax,ss, AUCinf, AUCτ,ss, Tmax, Tmax,ss, t½, CL/F, and Vd/F; for IN-C005, AUCinf, Tmax, Tmax,ss, Cmin,ss, t½, CL/F, Vd/F, Cav,ss, CLss/F, Vss/F, PTF (peak to trough fluctuation), and R (accumulation ratio)

[Pharmacodynamic Assessments]:

1. Single Dosing Group (Korean Subjects)

   * Intragastric pH

     * Percent (%) duration of pH ≥4 in 24 hrs
     * Mean pH
     * Median pH
     * Change in pH from baseline to post-dose (Δduration %, Δmean pH, Δmedian pH, etc.)
   * Serum gastrin level

     * AUEGlast
     * Gmax
     * Change in gastrin level from baseline to study treatment (1d, 8d, and 15d)(ΔAUEGlast, ΔGmax, etc.)
2. Multiple Dosing Group (Caucasian Subjects)

   * Intragastric pH

     * Percent (%) duration of pH ≥4 in 24 hrs
     * Mean pH
     * Median pH
     * Change in pH from baseline to post-single dose and post-multiple doses (Δduration %, Δmean pH, Δmedian pH, etc.)
   * Serum gastrin level

     * AUEGlast
     * Gmax
     * Change in gastrin level from baseline to 1d and 7d (ΔAUEGlast, ΔGmax, etc.)

[Safety Assessments] <Single Dosing Group (Korean Subjects) and Multiple Dosing Group (Caucasian Subjects)>

1. AEs will be monitored with observable/objective symptoms, etc.
2. Physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests

ELIGIBILITY:
Inclusion Criteria:

* [For single dosing group only] Healthy Korean male aged 19 to 50 years (inclusive) at the time of signing the informed consent form (ICF)
* [For multiple dosing group only] Healthy Caucasian male aged 19 to 50 years (inclusive) at the time of signing the ICF (Caucasian subject is defined as a European who was born in Europe, has the duration of residence outside of Europe less than 10 years, and both of whose parents and grandparents are European-born).
* Body mass index (BMI) of ≥ 18.0 and ≤ 28.0 kg/m2 with a body weight ≥ 55.0 kg at screening. (BMI (kg/m2) = weight (kg) / {height (m)}2)
* Subjects with negative result in serum Helicobacter pylori antibody test.
* Voluntary participation in the study after being fully informed of and understanding the study completely, and provides his written informed consent prior to screening procedure
* Subjects who are eligible for this study in the opinion of the investigator based on the results of physical examination, clinical laboratory tests, interview, etc.

Exclusion Criteria:

* History or current evidence of clinically significant disorder of hepatic, renal, nervous, respiratory, endocrine, hemato-oncologic, cardiovascular, urinary, and/or psychiatric system.
* History or current evidence of gastrointestinal disease that may affect the safety and PD assessment for study treatment (e.g., gastrointestinal ulcer, gastritis, gastric cramp, gastroesophageal reflux disease, and Crohn's disease) or a history of gastrointestinal surgery (except for simple appendectomy or herniotomy).
* History or current evidence of clinically significant hypersensitivity to drugs containing IN-C005 or any ingredient of proton pump inhibitors and other drugs (such as aspirin and antibiotics).
* Subjects with positive result on serology tests (for hepatitis B, human immunodeficiency virus [HIV], and hepatitis C).
* Subjects with blood level of total bilirubin, AST (GOT), or ALT (GPT) > 1.5 X upper limit of normal range(ULN) at procedures performed during the screening period including those performed additionally.
* Subjects with eGFR < 60 ml/min/1.73m2 during the screening period including those performed additionally.
* Systolic blood pressure (SBP) of < 90 mmHg or > 140 mmHg, diastolic blood pressure (DBP) of < 50 mmHg or > 95 mmHg, or pulse rate of < 45 beats/min or > 100 beats/min on vital signs as measured in sitting position after taking a rest for at least 5 minutes at screening.
* Subjects with anatomical disorder that precludes insertion and maintenance of intragastric pH meter catheter or is expected to be intolerable to insertion of intragastric pH meter catheter.
* History of drug abuse or positive response to drug abuse on urine drug screening test.
* Subjects who received any prescription drug or herbal medication within 2 weeks of or any over-the-counter (OTC) drug, dietary supplements, or vitamins within 1 week of scheduled first dose or subjects who are expected to receive such medication during the study. (Note: a subject may participate in the study at the discretion of the investigator, provided that the subject meets all the other criteria).
* Subjects who participated in any other clinical study or bioequivalence study and received investigational product within 6 months prior to the scheduled first dose.
* Subjects who have donated whole blood within 2 months prior to the scheduled first dose, or have donated blood components or received transfusion within a month prior to the scheduled first dose.
* Excessive caffeine intake (> 5 units/day), continued use of alcohol (> 21 units/week, 1 unit = 10 g of pure alcohol), or inability to stop drinking while hospitalized.
* Positive result for cotinine on urine drug screening test or inability to quit smoking throughout the study.
* Subjects who have taken grapefruit-containing foods during the period from 24 hours (hrs) before hospitalization to discharge, or are unable to avoid grapefruit-containing foods during this period.
* Subjects who are unable to avoid caffeine-containing foods (e.g., coffee, tea [red tea, green tee, etc.], soda, coffee milk, and nutritive tonic drink) during the period from 24 hrs before hospitalization to discharge.
* Subjects who are unable to use medically acceptable contraceptive methods throughout the study.

  ► Medically acceptable contraceptive methods include:

  ① Use of intrauterine device with a proven birth control failure rate by the spouse (or partner);

  ② Simultaneous use of (male or female) barrier method and spermicide; and

  ③ Surgical sterilization of the subject or his partner (e.g., vasectomy, salpingectomy, tubal ligation, or hysterectomy).
* Subjects who are determined ineligible for study participation by the investigator for other reasons such as clinical laboratory abnormalities.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Evaluation [Single Dosing Group (Korean Subjects), Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Cmax of IN-C005
Pharmacokinetic Evaluation [Single Dosing Group (Korean Subjects), Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  AUClast of IN-C005
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Cmax,ss of IN-C005
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  AUCtau,ss of IN-C005

SECONDARY OUTCOMES:
Pharmacokinetic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  AUClast of M1
Pharmacokinetic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  Cmax of M1
Pharmacokinetic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  AUCinf of IN-C005 and M1
Pharmacokinetic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  Tmax of IN-C005 and M1
Pharmacokinetic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  t½ of IN-C005 and M1
Pharmacokinetic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  CL/F of IN-C005 and M1
Pharmacokinetic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  Vd/F of IN-C005 and M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  AUClast of M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Cmax of M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Cmax,ss of M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  AUCinf of IN-C005 and M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  AUCtau,ss of M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Tmax of IN-C005 and M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Tmax,ss of IN-C005 and M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  t½ of IN-C005 and M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  CL/F of IN-C005 and M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Vd/F of IN-C005 and M1
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Cmin,ss of IN-C005
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Cav,ss of IN-C005
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  CLss/F of IN-C005
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  Vss/F of IN-C005
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  PTF (peak to trough fluctuation) of IN-C005
Pharmacokinetic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  R (accumulation ratio) of IN-C005
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Percent (%) duration of pH ≥ 4 in 24 hours
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Mean pH
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Median pH
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Change in pH from baseline to post-dose of Δduration %
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Change in pH from baseline to post-dose of Δmean pH
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Change in pH from baseline to post-dose of Δmedian pH
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  AUEGlast(Area under the concentration-time curve of serum gastrin from time zero to the last point of quantifiable concentration)
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  Gmax (Maximum plasma concentration of gastrin)
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  Change in gastrin level from baseline to 1d and 7d of ΔAUEGlast
Pharmacodynamic Evaluation [Single Dosing Group (Korean Subjects)] | Up to 48 hours
  Change in gastrin level from baseline to 1d and 7d of ΔGmax
Pharmacodynamic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Percent (%) duration of pH ≥ 4 in 24 hours
Pharmacodynamic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Mean pH
Pharmacodynamic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Median pH
Pharmacodynamic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Pre-dose(0h) up to 24 hours after IP administration in each period
  Change in pH from baseline to post-single dose and post-multiple dose (Δduration %, Δmean pH, Δmedian pH, etc)
Pharmacodynamic Evaluation [Multiple Dosing Group (Caucasian Subjects)] | Up to 48 hours
  AUEGlast(Area under the concentration-time curve of serum gastrin from time zero to the last point of quantifiable concentration)
Pharmacodynamic Evaluation [Multiple Dosing Group (Caucasian Subjects] | Up to 48 hours
  Gmax (Maximum plasma concentration of gastrin)
Pharmacodynamic Evaluation [Multiple Dosing Group (Caucasian Subjects] | Up to 48 hours
  Change in gastrin level from baseline to 1d and 7d of ΔAUEGlast
Pharmacodynamic Evaluation [Multiple Dosing Group (Caucasian Subjects] | Up to 48 hours
  Change in gastrin level from baseline to 1d and 7d of ΔGmax

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital, Clinical Trial Center
Locations (1):
- Seoul National University Hospital, Seoul, South Korea